CLINICAL TRIAL: NCT01562730
Title: Incremental Value of Signal Processed Surface Electrocardiography (IECG) for Detecting Ischemic Heart Disease: Comparison With Computed Tomography Coronary Angiography (CTCA)
Brief Title: Myovista iECG for Detecting Ischemic Heart Disease: Comparison With Computed Tomography Coronary Angiography
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cardiocentro Ticino (Other)
Collaborators: Meditrial SrL (Industry)
Responsible Party: Principal Investigator, Angelo Auricchio, Principal Investigator, Cardiocentro Ticino
Other Study IDs: HTL-01-11
Record Dates: First submitted 2012-03-22; First posted 2012-03-26 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Myocardial Ischemia; Coronary Disease; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases; iECG; 12 leads ECG
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Coronary Disease; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- No previous cardiovascular disease: Individuals without any history of cardiovascular disease
- Previous cardiovascular disease: Individuals with history of cardiovascular disease

SUMMARY:
Study evaluates the new technique MyoVista™ iECG sensitivity and ability to predict myocardial diseases, comparing iECG results with Computed Tomography Coronary Angiography findings

DETAILED DESCRIPTION:
Clinical need

Non-invasive identification of patients with coronary artery disease using a single, highly reliable technique is challenging. Computed tomography coronary angiography (CTCA) has emerged as a patient-friendly, accurate diagnostic tool. Compared to invasive coronary angiography, the sensitivity and specificity of CTCA for detecting significant coronary stenosis has been reported to be higher than 90%. Moreover, CTCA allows the detection of nonobstructive coronary plaques (CAPs). However, the advantage of CTCA is frequently reduced by significantly higher radiation exposure.

New MyoVista™ iECG technology

The MyoVista™ (Heart Test Laboratories Inc., Colleyville, TX, USA) is a novel electrocardiographic device. The clinical set up of MyoVista™ is identical to that of a traditional 12-lead ECG but it acquires and processes signal information in a way that permits much greater resolution of the electrical activity associated with the myocardium (iECG). This technology property of Heart Test Laboratories allows analysis of the entire myocardium and provides visual indicators and waveforms for clinical evaluation.

Study rationale

MyoVista™ technology has been so far validated in cohorts of Asian patients undergoing a clinically-indicated coronary angiography. These studies showed high positive and negative predictive values for identification of CAD. In addition, preliminary studies performed in the USA suggest a potential incremental value of iECG over routine surface ECG as a screening tool for detection of subclinical LV dysfunction and latent cardiovascular risk.

The aim of this prospective controlled evaluation is to assess

1. the sensitivity, specificity, and predictive value of MyoVista™ iECG in consecutive individuals without any history of cardiovascular disease undergoing a clinically indicated Computed Tomography Coronary Angiography (CTCA) in detecting Coronary Artery Plaque (CAP) and/or Coronary Artery Disease (CAD) (Group 1);
2. the sensitivity, specificity, and predictive value of MyoVista™ iECG in consecutive individuals with history of cardiovascular disease undergoing a clinically indicated CTCA in detecting the extent of CAP or CAD (Group 2);
3. whether MyoVista™ iECG abnormality is a better predictor of traditional risk factors to prevalence of CAP in individuals without history of cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* chest pain,
* shortness of breath,
* syncope or equivocal stress testing including exercise ECG,
* myocardial perfusion imaging, or stress echocardiography unable to exclude significant coronary artery disease.
* All patients will provide written and oral consent to CTCA.
* Patient agrees to participate and signs the informed consent

Exclusion Criteria:

* usually renal insufficiency (serum creatinine >120 mol/l),
* contraindications to the administration of iodinated contrast,
* pregnancy, acute coronary syndromes,
* and ventricular and/or supraventricular arrhythmias.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive individuals undergoing a clinically indicated Computed Tomography Coronary Angiography
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Comparison between Myovista iECG findings and CTCA (gold standard) results | one day
  Comparison of findings from the two methods will be made to demonstrate that Myovista iECG is equally effective as CTCA in predicting CAPs and/or CAD in individuals with or without history of cardiovascular disease, in terms of sensitivity, specificity and predictive value

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Auricchio, MD PhD FESC, Principal Investigator — Fondazione Cardiocentro Ticino
Locations (1):
- Fondazione Cardiocentro Ticino, Lugano, Switzerland

REFERENCES:
- [Background] Faletra FF, Klersy C, D'Angeli I, Penco M, Procaccini V, Pasotti E, Marcolongo A, Pedrazzini GB, De Castro S, Scappaticci M, Moccetti T, Auricchio A. Relation between coronary atherosclerotic plaques and traditional risk factors in people with no history of cardiovascular disease undergoing multi-detector computed coronary angiography. Heart. 2009 Aug;95(15):1265-72. doi: 10.1136/hrt.2009.167098. Epub 2009 Apr 29. PMID 19406736
- [Background] Henneman MM, Schuijf JD, van Werkhoven JM, Pundziute G, van der Wall EE, Jukema JW, Bax JJ. Multi-slice computed tomography coronary angiography for ruling out suspected coronary artery disease: what is the prevalence of a normal study in a general clinical population? Eur Heart J. 2008 Aug;29(16):2006-13. doi: 10.1093/eurheartj/ehn284. Epub 2008 Jun 23. PMID 18573865
- [Background] DeLong ER, DeLong DM, Clarke-Pearson DL. Comparing the areas under two or more correlated receiver operating characteristic curves: a nonparametric approach. Biometrics. 1988 Sep;44(3):837-45. PMID 3203132
- See also: Fondazione Cardiocentro Ticino — http://www.cardiocentro.org
- See also: Heart Test Laboratories Inc. — http://www.hearttestlabs.com